CLINICAL TRIAL: NCT04647890
Title: A Phase II, Randomised, Double Blind, Placebo-controlled Study of the Pharmacokinetics, Pharmacodynamic Effects, and Safety, of Oral FT011 in Participants With Diffuse Systemic Sclerosis
Brief Title: Effects of FT011 in Systemic Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Certa Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CER-FT011-SSc01
Record Dates: First submitted 2020-11-16; First posted 2020-12-01 (Actual); Results first posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Scleroderma, Systemic; Scleroderma, Diffuse; Sclerosis, Systemic
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse | interventions — FT011

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- FT011 200mg (Experimental): 200mg once daily for 12 weeks
  Interventions: Drug: FT011
- FT011 400mg (Experimental): 400mg once daily for 12 weeks
  Interventions: Drug: FT011
- Placebo (Placebo Comparator): Placebo once daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FT011 — Two x 100mg capsules once daily for 12 weeks
  Arms: FT011 200mg
Drug: FT011 — Two x 200mg capsules once daily for 12 weeks
  Arms: FT011 400mg
Drug: Placebo — Two placebo capsules once daily for 12 weeks
  Arms: Placebo

SUMMARY:
FT011 is an anti-fibrotic drug that is being tested as a treatment for scleroderma. This study is being conducted to see what the body does to the drug (pharmacokinetics), and what the drug does to the body (pharmacodynamics).

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to any study procedures and who agree to adhere to all protocol requirements.
2. Aged 18 to 75 years inclusive at the time of consent.
3. Have a classification of systemic sclerosis, as defined by American College of Rheumatology (ACR) and European League Against Rheumatism (EULAR) criteria with disease duration ≤10 years from first non-Raynaud phenomenon manifestation.
4. Have a diagnosis of diffuse cutaneous SSc defined as systemic sclerosis with skin thickening on the upper arms proximal to the elbows, on the upper legs proximal to the knees, or on the trunk.
5. Have skin thickening in a body area suitable for repeat biopsy.
6. Have a mRSS at Screening of ≥15 to ≤40.
7. FVC ≥50% of predicted at Screening.
8. If on azathioprine, mycophenolate mofetil, or hydroxychloroquine, have been on a stable dose for at least 2 months prior to baseline.
9. Women of childbearing potential (WOCPB) and males with partners of child-bearing potential must agree to use highly effective contraception (a failure rate of <1%), for the duration of the study and until three months after their last dose of IMP.

Exclusion Criteria:

1. Pregnant or breast-feeding, or plan to become pregnant during the study.
2. Have received any IMP within 30 days or 5 half-lives prior to randomisation (4 months if the previous drug was a new chemical entity), whichever is longer.
3. Have known or suspected contraindications to the IMP.
4. Have severe or unstable SSc or end-stage organ involvement as evidenced by:

   1. On an organ transplantation list or has received an organ transplant including autologous stem cell transplant.
   2. Renal crisis within 1 year prior to Baseline.
5. Interstitial lung disease or pulmonary hypertension requiring constant oxygen therapy. This excludes oxygen used to aid sleep or exercise.
6. Gastrointestinal dysmotility requiring total parenteral nutrition or requiring hospitalisation within the 6 months prior to Baseline.
7. Concomitant inflammatory myositis, rheumatoid arthritis, or systemic lupus erythematosus when definite classification criteria for those diseases are met (Bohan and Peter criteria for polymyositis and dermatomyositis)
8. SSc-like illnesses related to exposures or ingestions
9. The use of the following drugs within the specified periods:

   1. Methotrexate in the 2 weeks prior to Day 1
   2. Other anti-fibrotic agents including D-penicillamine or tyrosine kinase inhibitors (nilotinib, imatinib, dasatinib) in the month prior to Screening.
   3. Biologic drugs such as tumour necrosing factor (TNF) inhibitors, tocilizumab, or Janus kinase (JAK) inhibitors, in the 3 months prior to Screening.
   4. Rituximab in the 6 months prior to Screening.
   5. Cyclophosphamide oral or IV in the 3 months prior to Screening.
   6. Oral prednisolone >10 mg per day or IV steroids in the month prior to Screening.
10. Have any malignancy not considered cured (except basal cell or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix); a subject is considered cured if there has been no evidence of cancer recurrence for the 6 years prior to randomisation.
11. Have aspartate transaminase (AST), alanine transaminase (ALT), gamma-glutamyl transferase (GGT), lactate dehydrogenase (LDH), or bilirubin values above the upper limit of normal (ULN) at Screening or Baseline, or evidence of hepatic disease as determined by any one of the following: history of hepatic encephalopathy, history of oesophageal varices, or history of portacaval shunt.
12. Estimated glomerular filtration rate (eGFR) <60mL/min, urinary albumin/creatinine ratio >30mg/g.
13. Haemoglobin < 80 g/L, platelets < 90 x 109/L, or neutrophil count < 1.4 x 109/L
14. Other than SSc, have any other medical condition or significant co-morbidities, clinically relevant social or psychiatric conditions, or any finding during Screening, which in the investigator's opinion may put the subject at risk or interfere with the study objectives.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-07-19 (Actual); Primary Completion 2022-10-12 (Actual); Study Completion 2022-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Darren Kelly, PhD, Study Director — Certa Therapeutics Pty Ltd
Locations (10):
- Australia (2):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
- Certa SSc trial site, Nijmegen, Netherlands
- Poland (4):
  - Certa SSc trial site, Bydgoszcz
  - Certa SSc trial site, Krakow
  - Certa SSc trial site, Malbork
  - Certa SSc trial site, Warsaw
- Certa SSc trial site, Barcelona, Spain
- Ukraine (2):
  - Certa SSc trial site, Kyiv
  - Certa SSc trial site, Poltava

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | FT011 200mg | FT011 400mg | Placebo
Started | 10 | 10 | 10
Completed | 9 | 9 | 10
Not Completed | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FT011 200mg | FT011 400mg | Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 9 | 8 | 9 | 26
  >=65 years | 1 | 2 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 6 | 22
  Male | 3 | 1 | 4 | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 10 | 10 | 10 | 30
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: FT011 Levels in Plasma
Description: Measurement of maximum concentration (cmax) of FT011. First dose Cmax and last dose Cmax for each participant were averaged together to calculate a single mean Cmax for each treatment arm
Time Frame: Mean of cmax post first dose and cmax post last dose
Population: Placebo participants not tested
Measure: Mean (Standard Deviation); unit: ug/mL
Arm/Group | FT011 200mg | FT011 400mg | Placebo
Number analyzed (Participants) | 9 | 10 | 0
ug/mL | 5.45 (1.94) | 10.3 (4.27) |

2. Primary Outcome: FT011 Levels in Plasma
Description: Measurement of time to cmax (tmax). First dose tmax and last dose tmax for each participant were averaged together to calculate a single mean tmax for each treatment arm
Time Frame: Mean of time to cmax post first dose and time to cmax post last dose
Population: Placebo participants not tested
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | FT011 200mg | FT011 400mg | Placebo
Number analyzed (Participants) | 9 | 10 | 0
hours | 4.19 (1.75) | 4.20 (1.61) |

3. Primary Outcome: FT011 Levels in Plasma
Description: Measurement of area under the concentration time curve (AUC). First dose AUC and last dose AUC for each participant were averaged together to calculate a single mean AUC for each active arm
Time Frame: Mean of AUC hours post first dose and AUC hours post last dose
Population: Placebo participants not tested
Measure: Mean (Standard Deviation); unit: h*ug/mL
Arm/Group | FT011 200mg | FT011 400mg | Placebo
Number analyzed (Participants) | 9 | 10 | 0
h*ug/mL | 29.8 (11.1) | 57.8 (29.0) |

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) From Baseline to End of Study
Description: TEAEs per arm during study treatment and follow up periods
Time Frame: Baseline to Week 16
Measure: Count of Participants; unit: Participants
Arm/Group | FT011 200mg | FT011 400mg | Placebo
Number analyzed (Participants) | 10 | 10 | 10
Participants | 7 | 4 | 6

5. Secondary Outcome: mRSS Change From Baseline
Description: The mRSS is a validated physical evaluation of patient's skin thickness rated by clinical palpation using a 0-3 scale (0 = normal skin; 1 = mild thickness; 2 = moderate thickness; 3 = severe thickness with inability to pinch the skin into a fold) for each of 17 surface anatomic areas of the body: face, anterior chest, abdomen, and, with right and left sides of the body separately evaluated, the fingers, forearms, upper arms, thighs, lower legs, dorsum of hands and feet. Individual values are summed and defined as the total skin score. Total score is 0 to 51 with higher scores indicating worse symptomology
Time Frame: End of treatment (week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FT011 200mg | FT011 400mg | Placebo
Number analyzed (Participants) | 9 | 10 | 9
score on a scale | -3.7 (4.30) | -3.1 (4.15) | -2.7 (3.53)

6. Secondary Outcome: %FVC Change From Baseline
Description: Percent predicted FVC is calculated using equations incorporating age, gender, and race. It is calculated as (FVC Observed / FVC predicted) x 100, where FVC predicted is calculated relative to a reference population
Time Frame: End of treatment (Week 12)
Measure: Mean (Standard Deviation); unit: percentage of FVC change
Arm/Group | FT011 200mg | FT011 400mg | Placebo
Number analyzed (Participants) | 9 | 10 | 9
percentage of FVC change | -2 (2.24) | 4.7 (8.68) | -1.7 (4.24)

7. Secondary Outcome: Physician Global Assessment Change From Baseline
Description: The physician's assessment of the patient's SSc status will be scored on a 100-mm horizontal VAS, ranging from 0 on the extreme left end of the scale indicating "no disease activity" (symptom free), and 100 on the extreme right end indicating "worst imaginable disease activity".
Time Frame: End of treatment (Week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FT011 200mg | FT011 400mg | Placebo
Number analyzed (Participants) | 9 | 10 | 9
score on a scale | -15.2 (19.78) | -28.4 (22.89) | -6.3 (18.29)

8. Secondary Outcome: Patient Global Assessment Change From Baseline
Description: The Patient's Global Assessment represents the patient's overall assessment of current SSc status on a 100-mm horizontal VAS, ranging from 0 on the extreme left end of the scale indicating "no disease activity" (symptom free), and 100 on the extreme right end indicating "worst imaginable disease activity".
Time Frame: End of treatment (Week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FT011 200mg | FT011 400mg | Placebo
Number analyzed (Participants) | 9 | 10 | 9
score on a scale | 23 (9.53) | 10.8 (30.07) | 2.7 (19.99)

9. Secondary Outcome: Scleroderma HAQ-DI Change From Baseline
Description: The HAQ-DI consists of 20 questions referring to eight component sets consisting of dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Each item is scored from 0 to 3. The eight scores of the eight sections are summed and divided by 8. The total score indicates the patient's self-assessed level of disability - higher scores indicate worse symptomology. A negative change from baseline indicates improvement. The Scleroderma HAQ (SHAQ) includes an additional five scleroderma-specific visual analogue scales (VAS), addressing overall disease activity, Raynaud's phenomenon, finger ulcers, breathing, and intestinal problems. A composite VAS score is not created nor are the individual VAS scores incorporated into the HAQ DI score.
Time Frame: End of treatment (Week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FT011 200mg | FT011 400mg | Placebo
Number analyzed (Participants) | 9 | 10 | 9
score on a scale | -0.0694 (0.26598) | -0.2625 (0.23162) | 0.0278 (0.24826)

10. Secondary Outcome: Combined Response Index in Diffuse Cutaneous Systemic Sclerosis (CRISS) at Week 12
Description: CRISS components include modified Rodnan skin score (mRSS), forced vital capacity percent predicted (%FVC), Physician Global Assessment, Patient Global Assessment, and Health Assessment Questionnaire Disability-Index (HAQ-DI). The exponential algorithm determines the predicted probability of improvement from baseline, incorporating change in these 5 components. The outcome is a continuous variable between 0.0 and 1.0 (0 - 100%). A higher score indicates greater improvement
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FT011 200mg | FT011 400mg | Placebo
Number analyzed (Participants) | 9 | 10 | 8
score on a scale | 0.282 (0.4073) | 0.542 (0.4535) | 0.131 (0.2397)

11. Secondary Outcome: Scleroderma Clinical Trial Consortium Damage Index (SCTC-DI) Change From Baseline
Description: The SCTC-DI is a 23-item composite damage index to quantify organ damage in systemic sclerosis (0-55 scale; moderate damage >5, severe damage>12)
Time Frame: End of treatment (Week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FT011 200mg | FT011 400mg | Placebo
Number analyzed (Participants) | 9 | 10 | 9
score on a scale | -0.3 (0.71) | -0.3 (0.95) | -1.2 (2.54)

12. Secondary Outcome: 5-D Itch Scale Change From Baseline
Description: The 5-D itch scale is a 23-item validated instrument used to measure five domains of chronic itch: duration, degree, direction, disability, and distribution. Scores range from 5 to 25, with higher scores indicating a higher severity of chronic itch.
Time Frame: End of treatment (Week 12)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FT011 200mg | FT011 400mg | Placebo
Number analyzed (Participants) | 9 | 10 | 9
score on a scale | 0.7 (2.55) | -0.7 (4.47) | 0.2 (3.42)

ADVERSE EVENTS:
Time Frame: Over the duration of the study period (12 months)
Arm/Group | FT011 200mg | FT011 400mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 7/10 | 4/10 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FT011 200mg (N=10) | FT011 400mg (N=10) | Placebo (N=10)
Nasopharangytis (Infections and infestations) | 1 (1) | 2 (3) | 3 (3)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 2 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (2)
Genital candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Escherichia test positive (Investigations) | 0 (0) | 1 (1) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Tenosynovitis stenosans (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Vocal cord disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Raynaud's phenomenon (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2021-11-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT04647890/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT04647890/SAP_001.pdf